CLINICAL TRIAL: NCT06760273
Title: Extended Observational Study on the Long-term Impact of Tobramycin Inhalation Solution for Pseudomonas Aeruginosa Eradication in Patients With Bronchiectasis: The ERASE II Study
Brief Title: Long-term Impact of Inhaled Tobramycin for Pseudomonas Aeruginosa Eradication in Bronchiectasis (ERASE II)
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Professor, Huadong Hospital
Other Study IDs: 20230329-1
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Bronchiectasis Adult
Keywords: bronchiectasis; Pseudomonas Aeruginosa; Eradication; Long-term impact; Observational study
MeSH Terms: conditions — Bronchiectasis; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum, pseudomonas aeruginosa strains
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who successfully eradicate Pseudomonas aeruginosa in ERASE study: no intervention
  Interventions: Other: No Intervention: Observational Cohort
- Patients who were not successful in eradicating Pseudomonas aeruginosa in the ERASE Study: No intervention
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Observational study, no additional intervention

SUMMARY:
The ERASE II study is a prospective follow-up study designed to assess the long-term impact of successful eradication of Pseudomonas aeruginosa (PA) in patients with bronchiectasis. Building on the findings of the initial ERASE study, which evaluated the efficacy and safety of Tobramycin Inhalation Solution, ERASE II aims to determine whether successful PA eradication influences patient prognosis over an extended period.

The study will involve a total observation period of 36 months, consisting of the initial 9 months of the ERASE study followed by an additional 27 months of comprehensive follow-up. Key outcomes to be assessed include patients' quality of life, lung function, frequency of pulmonary exacerbations, frequency of hospitalization, and overall treatment costs. Additionally, the study will examine the timing and incidence of any potential reinfections with Pseudomonas aeruginosa.

DETAILED DESCRIPTION:
Individuals with bronchiectasis are particularly susceptible to infections from Pseudomonas aeruginosa (PA), which can become chronic and lead to increased mortality and disease severity. To address this critical issue, we have designed a multi-center, 2×2 factorial randomized, double-blind, placebo-controlled trial known as the ERASE study. This trial aims to evaluate the efficacy and safety of Tobramycin Inhalation Solution in the eradication of Pseudomonas aeruginosa in bronchiectasis patients with newly or firstly isolated PA.

Building upon the findings of the ERASE study, the ERASE II study seeks to investigate whether successful eradication of PA influences the long-term prognosis of patients after the completion of the randomized controlled trial. To achieve this, we plan to extend the observation period to a total of 36 months, comprising the initial 9 months of the ERASE study, followed by an additional 27 months of comprehensive follow-up.

This extended observation period will enable us to assess the long-term impact of eradication therapy on various clinical outcomes, including patients' quality of life, lung function, frequency of pulmonary exacerbations, frequency of hospitalization, and overall economic treatment costs. Additionally, we will evaluate the timing of any potential reinfections/relapse with Pseudomonas aeruginosa, thereby providing valuable insights into the long-term benefits of eradication strategies in patients with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* all patients who participate the ERSE study
* write the informed consent form.

Exclusion Criteria:

* patients who were lost of follow up in the ERASE study
* ineligible for inclusion at the discretion of the researcher for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have participate the ERASE study (NCT06093191)
Sampling Method: Non-Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients successfully eradicating PA in each group at 15 months, defined as a negative sputum culture of PA at 6, 9, 12, 15 months. | 15 months
  The sputum culture will be performed in each group at 6, 9, 12, and 15 months after randomization

SECONDARY OUTCOMES:
The proportion of patients with negative PA sputum cultures at 12 months following randomization, defined as a negative sputum culture of PA at 6, 9, and 12 months. | 12 months
  The sputum culture will be performed in each group at 6, 9, and 12 months after randomization
The proportion of patients with negative PA sputum cultures at 21 months following randomization, defined as a negative sputum culture of PA at 6, 9, 12, 15 and 21 months. | 21 months
  The sputum culture will be performed in each group at 6, 9, 12, 15 and 21 months after randomization
The proportion of patients with negative PA sputum cultures at 27 months following randomization, defined as a negative sputum culture of PA at 6, 9, 12, 15, 21 and 27 months. | 27 months
  The sputum culture will be performed in each group at 6, 9, 12, 15, 21 and 27 months after randomization
The proportion of patients with negative PA sputum cultures at 27 months following randomization, defined as a negative sputum culture of PA at 6, 9, 12, 15, 21, 27 and 36 months. | 36 months
  The sputum culture will be performed in each group at 6, 9, 12, 15, 21, 27 and 36 months after randomization
The differences in the frequency of pulmonary exacerbations of bronchiectasis at 12, 15, 21, 27, and 36 months following randomization. | 36 months
  The occurrences of pulmonary exacerbations will be documented during the follow-up period.
The differences in time to the first pulmonary exacerbation of bronchiectasis following randomization. | 36 months
  The occurrences of pulmonary exacerbations will be documented during the follow-up period.
The differences in the frequency of severe pulmonary exacerbations of bronchiectasis at 12, 15, 21, 27, and 36 months following randomization. | 36 months
  The occurrences of severe pulmonary exacerbations, defined as those requiring hospitalization, will be recorded during the follow-up period.
The differences in time to the first severe pulmonary exacerbation of bronchiectasis following randomization. | 36 months
  The occurrences of severe pulmonary exacerbations, defined as those requiring hospitalization, will be recorded during the follow-up period.
The changes in the QoL-B-RSS score from baseline in each group at 12, 15, 21, 27, and 36 months following randomization. | 36 months
  The QoL-B-RSS score will be recorded in each group at baseline, 12, 15, 21, 27, and 36 months following randomization. The Quality-of-Life-Bronchiectasis (QoL-B) questionnaire is a disease-specific survey designed for patients with bronchiectasis. The Respiratory Symptoms scale is a component of the QoL-B questionnaire, with a scale range from 0 to 100. Higher scores on this scale signify a better health status.
The changes in the SGRQ total score from baseline in each group at 12, 15, 21, 27, and 36 months following randomization. | 36 months
  The SGRQ total score will be recorded in each group at baseline, 12, 15, 21, 27, and 36 months following randomization. This questionnaire is structured into 3 main components: symptoms, activity and impacts.
  Scale range is 0-100, lower scores indicating better health status.
  Each component of the questionnaire is scored separately in three steps:
  i. The weights for all items with a positive responses are summed. ii. The weights for missed items are deducted from the maximum possible weight for each component. The weights for all missed items are deducted from the maximum possible weight for the Total score.
  iii. The score is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage The Total score is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing result as a percentage The Total score is calculated in similar way.
The changes of Euroqual-5 Dimensions questionnaire following randomization. | 36 months
  The (EQ-5D-5L) scale will be assessed at baseline, 12, 15, 21, 27, and 36 months following randomization.The Euroqual-5 Dimensions questionnaire (EQ-5D) consists of two parts: health state description and evaluation. In the description part, health status is measured across five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents rate their severity level for each dimension using a five-level (EQ-5D-5L) scale.
  In the evaluation part, respondents assess their overall health status using the visual analogue scale (EQ-VAS), which ranges from 0 to 100, with higher scores indicating a better health status.
  Health states defined by the EQ-5D-5L descriptive system are converted into index values. This facilitates the calculation of Quality-Adjusted Life Years (QALYs), which are used to inform economic evaluations of healthcare interventions, according to guidelines found at https://euroqol.org.
Daily Symptoms Measured by the bronchiectasis exacerbation and symptom tool (BEST) | 27
  Daily Symptoms were recorded by the bronchiectasis exacerbation and symptom tool (BEST)
Changes in forced expiratory volume in 1 second [FEV1] at 12, 21, 27 and 36 months compared with baseline | 36 months
  Changes in forced expiratory volume in 1 second [FEV1] at 12, 21, 27 and 36 months compared with baseline
Changes in forced vital capacity [FVC] at 12, 21, 27 and 36 months compared with baseline | 36 months
  Changes in forced vital capacity [FVC] at 12, 21, 27 and 36 months compared with baseline
Changes in forced expiratory flow at 25-75% of forced vital capacity at 12, 21, 27 and 36 months compared with baseline | 36 months
  Changes in forced expiratory flow at 25-75% of forced vital capacity at 12, 21, 27 and 36 months compared with baseline
The cost of hospitalization during the follow-up period | 36 months
  The cost of hospitalization during the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, PhD, Principal Investigator — Huadong Hospital affiliated with Fudan University
Locations (58):
- China (58):
  - Anhui Chest Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujiang
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Institute of Respiratory Diseases, Shenzhen, Guangdong
  - The Eighth Affiliated Hospital of Sun Yat-Sen University, Shenzhen, Guangdong
  - Affiliated Hospital, Guangdong Medical College, Zhanjiang, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hainan General Hospital, Hainan Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital,Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital, Nantong University, Nantong, Jiangsu
  - The Sixth People's Hospital of Nantong City, Nantong, Jiangsu
  - Suzhou Science and Technology Town Hospital, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shangrao People's Hospital, Shangrao, Jiangxi
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shangdong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - The Shanghai Fifth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai pulmonary hospital, Shanghai, Shanghai Municipality
  - Baoshan District Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Shanghai Eighth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo District People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First People's Hospital of Anning City Affiliated to Kunming University of Science and Technology, Anning, Yunnan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhengjiang University, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing City, Jiaxing, Zhejiang
  - The Second Hospital of Jiaxing City, Jiaxing, Zhejiang
  - Fenghua District People's Hospital of Ningbo City, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Conceicao M, Shteinberg M, Goeminne P, Altenburg J, Chalmers JD. Eradication treatment for Pseudomonas aeruginosa infection in adults with bronchiectasis: a systematic review and meta-analysis. Eur Respir Rev. 2024 Jan 31;33(171):230178. doi: 10.1183/16000617.0178-2023. Print 2024 Jan 31. PMID 38296344
- [Result] Gao YH, Lu HW, Zheng HZ, Cao C, Chu DJ, Fan H, Fan XY, Gu HY, Guan WJ, Jie ZJ, Jin Y, Li W, Li YP, Li YY, Liu L, Liu XD, Luo H, Lv XD, Mo WQ, Song YL, Wang DX, Wang LW, Wang CZ, Xie M, Zhang M, Zheng CX, Mao B, Chotirmall SH, Chalmers JD, Qu JM, Xu JF. A phase 4 multicentre, 2x2 factorial randomised, double-blind, placebo-controlled trial to investigate the efficacy and safety of tobramycin inhalation solution for Pseudomonas aeruginosa eradication in bronchiectasis: ERASE. ERJ Open Res. 2024 Feb 26;10(1):00938-2023. doi: 10.1183/23120541.00938-2023. eCollection 2024 Jan. PMID 38410702
- [Result] Hill AT, Sullivan AL, Chalmers JD, De Soyza A, Elborn SJ, Floto AR, Grillo L, Gruffydd-Jones K, Harvey A, Haworth CS, Hiscocks E, Hurst JR, Johnson C, Kelleher PW, Bedi P, Payne K, Saleh H, Screaton NJ, Smith M, Tunney M, Whitters D, Wilson R, Loebinger MR. British Thoracic Society Guideline for bronchiectasis in adults. Thorax. 2019 Jan;74(Suppl 1):1-69. doi: 10.1136/thoraxjnl-2018-212463. No abstract available. PMID 30545985
- [Result] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110
- See also: An extended observational study of the ERASE study — https://clinicaltrials.gov/study/NCT06093191?cond=Bronchiectasis&term=Jin-fu%20xu&page=2&rank=15